CLINICAL TRIAL: NCT04449939
Title: A Phase I, Open-label Study to Assess the Pharmacokinetics of KY1005 After Single Dose Administration by Subcutaneous and Intravenous Route in Healthy Volunteers
Brief Title: A Study of Subcutaneous KY1005 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymab Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY1005-CT04
Record Dates: First submitted 2020-06-15; First posted 2020-06-29 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Immune System Diseases
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Intervention Model Description: Single centre, open-label, single dose, parallel group study to investigate the PK, safety and tolerability of KY1005 after s.c. and i.v. administration, with i.v. KY1005 as a reference treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Single dose of KY1005 by i.v. infusion
  Interventions: Drug: KY1005
- Group 2 (Experimental): Single lower dose KY1005 by s.c. injection
  Interventions: Drug: KY1005
- Group 3 (Experimental): Single higher dose KY1005 by s.c. injections
  Interventions: Drug: KY1005

INTERVENTIONS:
Drug: KY1005 — A human anti-OX40 ligand monoclonal antibody

SUMMARY:
Single centre, open-label, single dose, parallel group study to investigate the PK, safety and tolerability of KY1005 after subcutaneous (s.c.) and intravenous (i.v.) administration, with i.v. KY1005 as a reference treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-45 years at screening
* Body weight 60-120 kg
* Body mass index (BMI) in the range 18.0-30.0 kg/m^2 (inclusive)
* Deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs and laboratory tests of blood and urine

Exclusion Criteria:

* Clinically relevant abnormal findings at the screening assessment; acute or chronic illness; clinically relevant abnormal medical history or concurrent medical condition; positive tests for hepatitis B, hepatitis C, Human Immunodeficiency Virus (HIV)
* Drug or alcohol abuse
* Use of over-the-counter medication (with the exception of paracetamol [acetaminophen]) during the 7 days before the first dose of trial medication, or prescribed medication during the 28 days before first dose of trial medication
* Participation in other clinical trials of unlicensed medicines within the 3 months or 5 half-lives, whichever is longer, before admission to this study
* Loss of more than 400 mL blood, within the previous 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) after infusion | Baseline to day 92
Time at which Cmax is observed after infusion (tmax) | Baseline to day 92
Area under the concentration time curve from time 0 to last observation (AUC 0-t) | Baseline to day 92
Area under the concentration time curve from time 0 to infinity (AUC0-inf) | Baseline to day 92
Systemic clearance after i.v. infusion (CL) | Baseline to day 92
Apparent systemic clearance after s.c. injection (CL/F) | Baseline to day 92
Volume of distribution during the terminal phase after i.v. infusion (Vz) | Baseline to day 92
Apparent volume of distribution after s.c. injection (Vz/F) | Baseline to day 92
Steady-state volume of distribution after i.v. infusion (Vss) | Baseline to day 92
Weight-normalised Vss and Vz | Baseline to day 92
Half-life t½ | Baseline to day 92
Dose-normalised Cmax (Cmax/D) following s.c. and i.v. administration | Baseline to day 92
Absolute bioavailability (F) calculated as the ratio of AUC0-inf/D after i.v. and s.c. infusion | Baseline to day 92
Dose-normalised AUC0-inf (AUC0-inf/D) following s.c. and i.v. administration | Baseline to day 92

SECONDARY OUTCOMES:
Occurrence of TEAE | Baseline to day 92
Occurrence of TESAE | Baseline to day 92
Occurrence of local injection site reactions | Baseline to day 92
Changes in blood pressure mmHg (as a measure of safety and tolerability) | Baseline to day 92
Changes in respiratory rate measured as breaths per minute (as a measure of safety and tolerability) | Baseline to day 92
Changes in heart rate bpm (as a measure of safety and tolerability) | Baseline to day 92
Changes in tympanic temperature °C (as a measure of safety and tolerability) | Baseline to day 92
Changes in electrocardiograms PR, QR, QRS and QT intervals (as a measure of safety and tolerability) | Baseline to day 92

OTHER OUTCOMES:
Serum anti-KY1005 antibody titres | Baseline to day 92
Incidence of anti-KY1005 antibodies | Baseline to day 92

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, MBBS JCPTGP MPhil, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom